CLINICAL TRIAL: NCT02112032
Title: Phase 1 Study of Anti-PD-1 Antibody MK-3475 and Peginterferon Alfa-2b for Advanced Melanoma
Brief Title: Treatment of Advanced Melanoma With MK-3475 and Peginterferon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hassane M. Zarour, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Melanoma Research Alliance (Other)
Responsible Party: Sponsor-Investigator, Hassane M. Zarour, MD, Professor of Medicine, Immunology, and Dermatology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-105
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-01

CONDITIONS: Melanoma
Keywords: melanoma; advanced
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; spartalizumab; Immunoglobulin G; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Level 1 (Experimental): MK-3475: 2 mg/kg every 3 weeks by intravenous infusion for up to 2 years Peginterferon alfa-2b: 1 µg/kg every week by subcutaneous injection for up to 2 years
  Interventions: Drug: MK-3475; Drug: Peginterferon alfa-2b
- Dose Level 2 (Experimental): MK-3475: 2 mg/kg every 3 weeks by intravenous infusion for up to 2 years Peginterferon alfa-2b: 2 µg/kg every week by subcutaneous injection for up to 2 years
  Interventions: Drug: MK-3475; Drug: Peginterferon alfa-2b
- Dose Level 3 (Experimental): MK-3475: 2 mg/kg every 3 weeks by intravenous infusion for up to 2 years Peginterferon alfa-2b: 3 µg/kg every week by subcutaneous injection for up to 2 years
  Interventions: Drug: MK-3475; Drug: Peginterferon alfa-2b

INTERVENTIONS:
Drug: MK-3475 — This is a dose escalation study to determine the serious and non-serious adverse events that occur as the dose increases.
  Other Names: Anti-PD-1; SCH 900475; 1374853-91-4; Humanized X PD-1_mAb (H409A11) IgG4
Drug: Peginterferon alfa-2b — This is a dose escalation study to determine the serious and non-serious adverse events that occur from the combination of Peginterferon and MK-3475 as the doses increase.
  Other Names: Sylatron; 215647-85-1; Pegintron

SUMMARY:
This study is to test how safe it is to give the combination of PEG IFN-α2b (SYLATRON) and MK-3475, an investigational drug, to patients with advanced melanoma. Its effectiveness against melanoma will also be evaluated.

DETAILED DESCRIPTION:
This is a safety and dose-seeking study of combination MK-3475 and peginterferon alfa-2b for adult patients (≥18) with advanced melanoma. A total of 32 patients will be included. Subjects will undergo screening evaluations to determine eligibility within 28 days (4 weeks) of the first dose. Each 21 day dosing period will constitute a cycle.

Peginterferon alfa-2b is given subcutaneously, weekly according to the regimen below. peginterferon alfa-2b (Sylatron) is FDA-approved for the adjuvant treatment of patients with melanoma with microscopic or gross nodal involvement within 84 days of definitive surgical resection including complete lymphadenectomy.

MK-3475 is a potent humanized IgG4 mAb with high specificity of binding to the PD-1 receptor, thus inhibiting its interaction with PD-L1 and PD-L2. MK-3475 has an acceptable preclinical safety profile and is being advanced for clinical development as an immunotherapy for advanced malignancies. In this protocol, MK-3475 is being evaluated at 2 mg/kg intravenously every 3 weeks for 2 years in combination with peginterferon alfa-2b at 1 µg/kg/week, 2 µg/kg/week, or 3 µg/kg/week by subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically or cytologically confirmed diagnosis of unresectable stage III or IV melanoma. Patient may not have a diagnosis of uveal melanoma.
* Patients may be previously untreated or have received up to 3 prior systemic therapies for metastatic disease. Prior radiation therapy (any number) and interferon use in the adjuvant or metastatic disease settings is permitted (in this trial interferon is mainly used to enhance or initiate immune responses to MK-3475). Vaccine therapy will not be counted as systemic therapy. All prior therapies must have been discontinued for at least 4 weeks. A 2 week washout for kinase inhibitors is acceptable.
* Patients can be either ipilimumab naïve or refractory to ipilimumab, defined as received at least two doses of ipilimumab and documented disease progression. Patients who were re-treated with ipilimumab and patients who were on maintenance ipilimumab will be allowed to enter the trial as long as there is documented PD. Progressive disease will be defined as increase in tumor burden > 25% relative to nadir (minimum recorded tumor burden) which is confirmed by repeat assessment no less than four weeks from the date of the first documented PD. Once PD is confirmed, initial date of PD documentation will be considered as the date of disease progression.
* Full resolution of ipilimumab related AEs to baseline (including irAEs) off of steroid treatment (> 10 mg/day prednisone or equivalent dose) for irAEs for at least two weeks prior to first dose of study drug.

  1. No history of severe irAEs from ipilimumab of CTCAE Grade 4 requiring steroid treatment; no history of CTCAE Grade 3 requiring steroid treatment (> 10mg/day prednisone or equivalent dose) for > 12 weeks.
  2. Minimum of four weeks (wash out period) from the last dose of ipilimumab.
* Patients must consent to participate in the correlative studies and should have available tumor tissue for tumor biopsies.
* Patient must have measurable disease as per RECIST version 1.1. At least 1 of the tumor sites must be amenable to biopsy and this may not be the site of disease used to measure antitumor response.
* Patient is ≥ 18 years of age on day of signing informed consent.
* Patient must have a performance status of 0 or 1 on the ECOG Performance Scale
* Patient must have adequate organ function as indicated by the following laboratory values (within 4 weeks prior to starting the study drugs):

  1. Absolute neutrophil count (ANC) ≥ 1,500/uL
  2. Platelets ≥ 100,000/uL
  3. Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
  4. Serum creatinine ≤ 1.5 X upper limit of normal (ULN)
  5. Serum total bilirubin ≤ 1.5 X ULN OR direct bilirubin ≤ ULN for patients with total bilirubin level 1.5 ULN
  6. AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for patients with liver metastases
  7. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 X ULN unless the patient is receiving anticoagulant therapy
  8. Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless the patient is receiving anticoagulant therapy
* Patient has voluntarily agreed to participate by giving written informed consent/assent for the trial.
* Female patient of childbearing potential has a negative urine or serum pregnancy test within 7 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the patient to be eligible.
* Female patients enrolled in the study, who are not free from menses for > 2 years, post hysterectomy/oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy, or to abstain from heterosexual activity throughout the study, starting with the first dose of study drug at visit 1 through 120 days after the last dose of study drug. Approved contraceptive methods include for example: intra-uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception. Male patients must agree to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

* Patient who has had chemotherapy, radioactive, or biological cancer therapy within four weeks prior to the first dose of study drug, or who has not recovered to CTCAE Grade 1 or better from the AEs due to cancer therapeutics administered more than four weeks earlier. Subjects with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study.

Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

Note: Toxicity that has not recovered to ≤ Grade 1 is allowed if it meets the inclusion requirements for laboratory parameters defined in Inclusion Criterion #9.

* Patient is currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of study drug.
* Patient is expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Patient is on chronic systemic steroid therapy (> 10 mg/kg prednisone or equivalent) within two weeks before the planned date for first dose randomized treatment or on any other form of immunosuppressive medication (Premedication with corticosteroid for nausea is permitted.)
* Patient has a known history of a hematologic malignancy, primary brain tumor or sarcoma, or of another primary solid tumor, unless the patient has undergone potentially curative therapy with no evidence of that disease for five years.

Note: The time requirement also does not apply to patients who underwent successful definitive resection of basal or squamous cell carcinoma of the skin, superficial bladder cancer, in situ cancers including cervical cancer, breast cancer, melanoma, or other in situ cancers.

* Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by MRI for at least four weeks prior to the first dose of study drug), have no evidence of new or enlarging brain metastases and are off systemic steroids (≤ 10 mg/day prednisone or equivalent) for at least two weeks prior to enrollment.
* Patient previously had a severe hypersensitivity reaction to treatment with another mAb or IFN-α2b.
* Patient has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo, type I diabetes, resolved childhood asthma/atopy would be exceptions to this rule. Patients who require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients with hypothyroidism stable on hormone replacement will also not be excluded from the study.
* Patient has evidence of interstitial lung disease.
* Serious illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), bleeding disorders, autoimmune diseases, severe obstructive or restrictive pulmonary diseases, active systemic infections, and inflammatory bowel disorders. This includes HIV or AIDS-related illness, or active HBV and HCV.
* Patient had prior treatment with any other anti-PD-1, or PD-L1 or PD-L2 agent.
* Patient has an active infection requiring systemic therapy.
* Patient has known history of human Immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Patient positive for Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA [qualitative] is detected).
* Patient has received a live vaccine within 4 weeks prior to the first dose of treatment.
* Patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patient is, at the time of signing informed consent, a regular user (including illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
* Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Patient has prior history of intolerance to adjuvant interferon-α therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | 29 days

SECONDARY OUTCOMES:
Time to Disease Progression | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hassane Zarour, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No